CLINICAL TRIAL: NCT03875235
Title: A Phase III Randomized, Double-Blind Placebo Controlled, Multi-Regional, International Study of Durvalumab in Combination With Gemcitabine Plus Cisplatin Versus Placebo in Combination With Gemcitabine Plus Cisplatin for Patients With First-Line Advanced Biliary Tract Cancers
Brief Title: Durvalumab or Placebo in Combination With Gemcitabine/Cisplatin in Patients With 1st Line Advanced Biliary Tract Cancer (TOPAZ-1)
Acronym: TOPAZ-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D933AC00001; 2023-507405-34-00 (Registry Identifier: CTIS (EU)); 2018-004688-30 (EudraCT Number)
Record Dates: First submitted 2019-03-13; First posted 2019-03-14 (Actual); Results first posted 2023-04-13 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Biliary Tract Neoplasms
Keywords: First-Line Advanced Biliary Tract Cancers (BTC); Durvalumab; Gemcitabine/Cisplatin; Placebo
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: Durvalumab in Combination with Gemcitabine plus Cisplatin Placebo in Combination with Gemcitabine plus Cisplatin
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Durvalumab + Gemcitabine + Cisplatin
  Interventions: Drug: Durvalumab
- Placebo Arm (Placebo Comparator): Placebo + Gemcitabine + Cisplatin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Durvalumab — IV infusion every 3 weeks with gemcitabine plus cisplatin up to 8 cycles followed by monotherapy every 4 weeks until disease progression or other discontinuation criteria.
  Arms: Treatment Arm
Drug: Placebo — IV infusion every 3 weeks with gemcitabine plus cisplatin up to 8 cycles followed by monotherapy every 4 weeks until disease progression or other discontinuation criteria.
  Arms: Placebo Arm

SUMMARY:
Durvalumab or Placebo in Combination With Gemcitabine/Cisplatin in Patients With 1st Line Advanced Biliary Tract Cancer (TOPAZ-1)

DETAILED DESCRIPTION:
A Phase III Randomized, Double-Blind Placebo Controlled, Multi-Regional, International Study of Durvalumab in Combination with Gemcitabine Plus Cisplatin Versus Placebo in Combination with Gemcitabine Plus Cisplatin for Patients With First-Line Advanced Biliary Tract Cancers.

ELIGIBILITY:
Inclusion

1. Histologically confirmed, unresectable advanced or metastatic biliary tract, including cholangiocarcinoma (intrahepatic or extrahepatic) and gallbladder carcinoma.
2. Patients with previously untreated disease if unresectable or metastatic at initial diagnosis will be eligible.
3. Patient with recurrent disease >6 months after curative surgery or >6 months after the completion of adjuvant therapy (chemotherapy and/or radiation) will be eligible.
4. WHO/ECOG PS of 0 or 1

Exclusion

1. History of another primary malignancy
2. Brain metastases or spinal cord compression
3. Uncontrolled intercurrent illness
4. Major surgical procedure within 28 days prior to the first dose of IP.
5. Prior locoregional therapy such as radioembolization

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 810 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Cohen, Study Director — AstraZeneca
Locations (106):
- United States (15):
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Fort Myers, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Westwood, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Burlington, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Seattle, Washington
- Argentina (5):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Rosario
  - Research Site, San Salvador de Jujuy
- Bulgaria (3):
  - Research Site, Burgas
  - Research Site, Sofia
  - Research Site, Varna
- Chile (2):
  - Research Site, Santiago
  - Research Site, Temuco
- China (19):
  - Research Site, Baoding
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Chongqing
  - Research Site, Foshan
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Suzhou
  - Research Site, Xi'an
  - Research Site, Zhengzhou
  - Research Site, Zhuhai
- France (7):
  - Research Site, Clichy
  - Research Site, Dijon
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Poitiers
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Kowloon
- India (4):
  - Research Site, Gūrgaon
  - Research Site, Kolkata
  - Research Site, Mumbai
  - Research Site, New Delhi
- Italy (6):
  - Research Site, Faenza
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Roma
  - Research Site, Verona
- Japan (8):
  - Research Site, Chūōku
  - Research Site, Kashiwa
  - Research Site, Kitaadachi-gun
  - Research Site, Mitaka-shi
  - Research Site, Osaka
  - Research Site, Suita-shi
  - Research Site, Wakayama
  - Research Site, Yokohama
- Poland (6):
  - Research Site, Gdansk
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Russia (5):
  - Research Site, Barnaul
  - Research Site, Kostroma
  - Research Site, Moscow
  - Research Site, Omsk
  - Research Site, Saint Petersburg
- South Korea (2):
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Taiwan (6):
  - Research Site, Chiayi City
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (5):
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Muang
  - Research Site, Si Sa Ket
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Mersin
- United Kingdom (7):
  - Research Site, Bristol
  - Research Site, Cambridge
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Oxford
  - Research Site, Romford
  - Research Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Antonuzzo L, Takahashi H, Park JO, Sookprasert A, Gillmore R, Yang SS, Cundom J, Petrova M, Vaccaro G, Holmblad M, Zotkiewicz M, Wang J, Rokutanda N, Oh DY. Immune-mediated adverse events in the randomized phase 3 TOPAZ-1 study of durvalumab plus gemcitabine and cisplatin in advanced biliary tract cancer. Oncologist. 2025 Jul 4;30(7):oyaf148. doi: 10.1093/oncolo/oyaf148. PMID 40622010
- [Derived] Oh DY, He AR, Qin S, Chen LT, Okusaka T, Kim JW, Suksombooncharoen T, Lee MA, Kitano M, Burris HA, Bouattour M, Tanasanvimon S, Zaucha R, Avallone A, Cundom J, Kuzko A, Wang J, Xynos I, Vogel A, Valle JW. Durvalumab plus chemotherapy in advanced biliary tract cancer: 3-year overall survival update from the phase III TOPAZ-1 study. J Hepatol. 2025 Nov;83(5):1092-1101. doi: 10.1016/j.jhep.2025.05.003. Epub 2025 May 15. PMID 40381735
- [Derived] Oh DY, He AR, Bouattour M, Okusaka T, Qin S, Chen LT, Kitano M, Lee CK, Kim JW, Chen MH, Suksombooncharoen T, Ikeda M, Lee MA, Chen JS, Potemski P, Burris HA 3rd, Ostwal V, Tanasanvimon S, Morizane C, Zaucha RE, McNamara MG, Avallone A, Cundom JE, Breder V, Tan B, Shimizu S, Tougeron D, Evesque L, Petrova M, Zhen DB, Gillmore R, Gupta VG, Dayyani F, Park JO, Buchschacher GL Jr, Rey F, Kim H, Wang J, Morgan C, Rokutanda N, Zotkiewicz M, Vogel A, Valle JW. Durvalumab or placebo plus gemcitabine and cisplatin in participants with advanced biliary tract cancer (TOPAZ-1): updated overall survival from a randomised phase 3 study. Lancet Gastroenterol Hepatol. 2024 Aug;9(8):694-704. doi: 10.1016/S2468-1253(24)00095-5. Epub 2024 May 29. PMID 38823398
- [Derived] Keller HR, Fluke L, Forrester JA, Wolf RF. Identifying Indications for Neoadjuvant Therapy in Cholangiocarcinoma. Oncology (Williston Park). 2024 Apr 11;38(4):160-162. doi: 10.46883/2024.25921017. PMID 38661512
- [Derived] Oh DY, Ruth He A, Qin S, Chen LT, Okusaka T, Vogel A, Kim JW, Suksombooncharoen T, Ah Lee M, Kitano M, Burris H, Bouattour M, Tanasanvimon S, McNamara MG, Zaucha R, Avallone A, Tan B, Cundom J, Lee CK, Takahashi H, Ikeda M, Chen JS, Wang J, Makowsky M, Rokutanda N, He P, Kurland JF, Cohen G, Valle JW. Durvalumab plus Gemcitabine and Cisplatin in Advanced Biliary Tract Cancer. NEJM Evid. 2022 Aug;1(8):EVIDoa2200015. doi: 10.1056/EVIDoa2200015. Epub 2022 Jun 1. PMID 38319896
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933AC00001&attachmentIdentifier=f0f0274f-a72a-4d83-8200-e6a74d44d8fe&fileName=D933AC00001_-___Statistical_Analysis_Plan-redact.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933AC00001&attachmentIdentifier=88a80119-302b-4810-bce2-623ab0a77f31&fileName=d933ac00001-oncology-late-phase-master-csp-v8-redact.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933AC00001&attachmentIdentifier=7f0ef0d5-6fe8-4acc-8de5-143b4c68c4d9&fileName=d933ac00001-study-synopsis-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study is active, not recruiting and conducted in 17 countries with 685 patients who were randomized prior to or on 18 December 2020. Results are reported for the study at data cut-off (DCO) 11 August 2021.
Pre-assignment Details: Eligible patients previously untreated for unresectable locally advanced or metastatic Biliary Tract Cancer (BTC) were randomized in a 1:1 ratio with either Durvalumab in combination with Gemcitabine/Cisplatin or Placebo in combination with Gemcitabine/Cisplatin. Randomization was stratified by disease status (initially unresectable versus recurrent) and primary tumor site (IHCC versus EHCC versus GBC).
Groups:
- Durvalumab + Gemcitabine + Cisplatin: Drug: Durvalumab IV infusion every 3 weeks with gemcitabine plus cisplatin up to 8 cycles followed by monotherapy every 4 weeks until disease progression or other discontinuation criteria.
- Placebo + Gemcitabine + Cisplatin: Drug: Placebo IV infusion every 3 weeks with gemcitabine plus cisplatin up to 8 cycles followed by monotherapy every 4 weeks until disease progression or other discontinuation criteria.
Period: Overall Study
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Placebo + Gemcitabine + Cisplatin
Started | 341 | 344
Treated | 338 | 342
Completed | 0 | 0
Not Completed | 341 | 344
Not completed — Ongoing study treatment | 63 | 20
Not completed — Off treatment | 77 | 91
Not completed — Withdrawal by Subject | 3 | 10
Not completed — Death | 198 | 223

BASELINE CHARACTERISTICS:
Population: Baseline analysis was based on all patients in the full analysis set (FAS), which comprised all patients randomized prior to or on 18 December 2020. Patients were included in the analysis in the treatment arm to which they were randomized, regardless of the treatment they received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Placebo + Gemcitabine + Cisplatin | Total
Number analyzed (Participants) | 341 | 344 | 685
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.2 (10.49) | 62.6 (10.66) | 62.4 (10.57)
Age, Customized [Count of Participants; unit: Participants]
  Age group (years): < 65 years | 181 | 184 | 365
  Age group (years): >=65 - < 75 years | 122 | 114 | 236
  Age group (years): >= 75 years | 38 | 46 | 84
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 168 | 340
  Male | 169 | 176 | 345
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian of Alaska Native | 0 | 1 | 1
  Race: Asian | 185 | 201 | 386
  Race: Black or African American | 8 | 6 | 14
  Race: White | 131 | 124 | 255
  Race: Other | 17 | 12 | 29

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time from the date of randomization until death due to any cause. Any patient not known to have died at the time of analysis was censored based on the last recorded date on which the patient was known to be alive. Median OS was calculated using the Kaplan-Meier technique. The second interim analysis was pre-specified after approximately 397 OS events occurred in both arms (59% maturity).
Time Frame: From date of randomization until death due to any cause. Assessed up to maximum of approximately 27 months (from date of randomization to primary analysis data cut-off)
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 341 | 344
Months | 12.8 [11.1 to 14.0] | 11.5 [10.1 to 12.5]
Statistical Analysis 1: Comparison: Durvalumab + Gemcitabine + Cisplatin vs Placebo + Gemcitabine + Cisplatin; The 2-sided significance level for OS at the second interim analysis was 3%; Test type: Superiority; p = 0.021, Log Rank — The analysis was performed using a stratified log-rank test adjusting for disease status (initially unresectable versus recurrent) and primary tumor location (IHCC versus EHCC versus GBC), and tested at 0.03 significance level; Hazard Ratio (HR) = 0.80, 97% CI 2-sided [0.64 to 0.99] — The HR and CI were estimated from a stratified Cox proportional hazard model adjusting for disease status and primary tumor location; 95% CI 0.66 to 0.97

2. Primary Outcome: Overall Survival (OS) Rate at 18 Months
Description: as for outcome 1
Time Frame: From date of randomization until death due to any cause. Calculated at 18 months using the Kaplan-Meier technique.
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 341 | 344
Percentage of Participants | 35.1 [29.1 to 41.2] | 25.6 [19.9 to 31.7]

3. Primary Outcome: Overall Survival (OS) Rate at 24 Months
Description: as for outcome 1
Time Frame: From date of randomization until death due to any cause. Calculated at 24 months using the Kaplan-Meier technique.
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 341 | 344
Percentage of Participants | 24.9 [17.9 to 32.5] | 10.4 [4.7 to 18.8]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS based on investigator assessments according to RECIST version 1.1 was defined as time from date of randomization until date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the patient withdrew from randomized therapy or received another anticancer therapy prior to progression. Progression (i.e., PD) was defined as at least a 20% increase in the sum of diameters of target lesions (TLs) and an absolute increase of ≥5mm, taking as reference the smallest sum of diameters since treatment started including the baseline sum of diameters, or a measurable increase in a non-target lesion, or the appearance of new lesions. Median PFS was calculated using the Kaplan-Meier technique.
Time Frame: Tumor assessments every 6 weeks after randomization for the first 24 weeks and then every 8 weeks thereafter until date of RECIST 1.1 defined radiological progressive disease or death. Assessed up to maximum of approximately 27 months.
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 341 | 344
Months | 7.2 [6.7 to 7.4] | 5.7 [5.6 to 6.7]
Statistical Analysis 1: Comparison: Durvalumab + Gemcitabine + Cisplatin vs Placebo + Gemcitabine + Cisplatin; The 2-sided significance level for PFS at the second interim analysis was 4.81%; Test type: Superiority; p = 0.001, Log Rank — The p-value is based on a stratified log-rank test adjusting for disease status (initially unresectable versus recurrent) and primary tumor location (IHCC versus EHCC versus GBC), and tested at 0.0481 significance level; Hazard Ratio (HR) = 0.75, 95.19% CI 2-sided [0.63 to 0.89] — [estimate comment as in outcome 1, analysis 1]; 95% CI 0.63 to 0.89

5. Secondary Outcome: Progression-free Survival (PFS) Rate at 9 Months
Description: as for outcome 4
Time Frame: Tumor assessments every 6 weeks after randomization for the first 24 weeks and then every 8 weeks thereafter until date of RECIST 1.1 defined radiological progressive disease or death. Calculated at 9 months using the Kaplan-Meier technique.
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 341 | 344
Percentage of Participants | 34.8 [29.6 to 40.0] | 24.6 [20.0 to 29.5]

6. Secondary Outcome: Progression-free Survival (PFS) Rate at 12 Months
Description: as for outcome 4
Time Frame: Tumor assessments every 6 weeks after randomization for the first 24 weeks and then every 8 weeks thereafter until date of RECIST 1.1 defined radiological progressive disease or death. Calculated at 12 months using the Kaplan-Meier technique
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 341 | 344
Percentage of Participants | 16.0 [12.0 to 20.6] | 6.6 [4.1 to 9.9]

7. Secondary Outcome: Objective Response Rate (ORR)
Description: Disease assessments based on investigator assessments were determined by using RECIST version 1.1 guidelines. The ORR was defined as the percentage of patients with confirmed complete response (CR) or confirmed partial response (PR). The CR was defined as disappearance of all target and non-target lesions and no new lesions. The PR was defined as >= 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new non-target lesion. A confirmed CR or PR was defined as 2 CRs or 2 PRs with no evidence of progression in-between. Patients who discontinued randomized treatment without progression, received a subsequent anti-cancer therapy and then responded were not included as responders for ORR.
Time Frame: Tumor assessments (per RECIST 1.1) every 6 weeks for the first 24 weeks relative to the date of randomization and then every 8 weeks thereafter. Assessed up to maximum of approximately 27 months.
Population: Full analysis set - subjects with measurable disease at baseline
Measure: Number; unit: Percentage of Participants
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 341 | 343
Percentage of Participants | 26.7 | 18.7
Statistical Analysis 1: Comparison: Durvalumab + Gemcitabine + Cisplatin vs Placebo + Gemcitabine + Cisplatin; Test type: Superiority; p = 0.011, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.60, 95% CI 2-sided [1.11 to 2.31] — OR and CI were estimated from a stratified CMH test adjusting for disease status and primary tumor location

8. Secondary Outcome: Duration of Response (DoR)
Description: The DoR was defined as the time from the date of first documented OR (confirmed CR or confirmed PR) until date of documented progression (PD) based on investigator assessments by using RECIST version 1.1 or death in absence of disease progression (i.e. date of PFS event or censoring - date of first response + 1) . A confirmed CR was defined in above outcome measures. The PD was defined at least 20% increase in sum of diameters of target lesions (compared with nadir at 2 consecutive visits with an absolute increase of 5 mm), unequivocal progression of existing non-target lesions or new lesion. For participants who were alive and no documented PD at the time of data cutoff for analysis, DoR was censored at the last evaluable disease assessment date. Median DoR was calculated using Kaplan-Meier method.
Time Frame: Tumor assessments (per RECIST 1.1) every 6 weeks for first 24 weeks relative to the date of randomization and then every 8 weeks thereafter. Assessed up to maximum of approximately 27 months.
Population: Full analysis set - subjects with objective response and measurable disease at baseline
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 91 | 64
Months | 6.4 [5.9 to 8.1] | 6.2 [4.4 to 7.3]

9. Secondary Outcome: Duration of Response (DoR): Percentage Remaining in Response at 9 Months
Description: as for outcome 8
Time Frame: Tumor assessments (per RECIST 1.1) every 6 weeks for first 24 weeks relative to the date of randomization and then every 8 weeks thereafter. Calculated at 9 months using the Kaplan-Meier technique
Population: Full analysis set - subjects with objective response and measurable disease at baseline
Measure: Number; unit: Percentage of Participants
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 91 | 64
Percentage of Participants | 32.6 | 25.3

10. Secondary Outcome: Duration of Response (DoR): Percentage Remaining in Response at 12 Months
Description: as for outcome 8
Time Frame: Tumor assessments (per RECIST 1.1) every 6 weeks for first 24 weeks relative to the date of randomization and then every 8 weeks thereafter. Calculated at 12 months using the Kaplan-Meier technique
Population: Full analysis set - subjects with objective response and measurable disease at baseline
Measure: Number; unit: Percentage of Participants
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 91 | 64
Percentage of Participants | 26.1 | 15.0

11. Secondary Outcome: Disease Control Rate (DCR) - Overall
Description: Disease control rate based on investigator assessments according to RECIST version 1.1 was defined as the rate of best objective response of complete response (CR), partial response (PR) or stable disease (SD).
Time Frame: as for outcome 7
Population: Full analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 341 | 344
Percentage of Participants | 85.3 | 82.6

12. Secondary Outcome: Disease Control Rate (DCR) - 24 Weeks
Description: Disease control rate based on investigator assessments according to RECIST version 1.1 was defined as the rate of best objective response of complete response (CR) or partial response (PR) by week 24 or who have stable disease (SD) at least 24 weeks following start of treatment.
Time Frame: Tumor assessments (per RECIST 1.1) every 6 weeks for the first 24 weeks relative to the date of randomization.
Population: Full analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 341 | 344
Percentage of Participants | 57.5 | 48.3

13. Secondary Outcome: Disease Control Rate (DCR) - 32 Weeks
Description: Disease control rate based on investigator assessments according to RECIST version 1.1 was defined as the rate of best objective response of complete response (CR) or partial response (PR) by week 32 or who have stable disease (SD) at least 32 weeks following start of treatment.
Time Frame: Tumor assessments (per RECIST 1.1) every 6 weeks for the first 24 weeks relative to the date of randomization and then every 8 weeks thereafter.
Population: Full analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 341 | 344
Percentage of Participants | 41.9 | 36.3

14. Secondary Outcome: Disease Control Rate (DCR) - 48 Weeks
Description: Disease control rate based on investigator assessments according to RECIST version 1.1 was defined as the rate of best objective response of complete response (CR) or partial response (PR) by week 48 or who have stable disease (SD) at least 48 weeks following start of treatment.
Time Frame: as for outcome 13
Population: Full analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 341 | 344
Percentage of Participants | 35.2 | 27.0

ADVERSE EVENTS:
Time Frame: Adverse events: from first dose of study medication up to 90 days after the last dose of study medication or until the initiation of the first subsequent therapy (whichever comes first), up to maximum of approximately 27 months. All-cause mortality (death due to any cause): from randomization up to analysis DCO (11 August 2021). Maximum timeframe of approximately 27 months.
Description: There were 341 patients randomized to Durvalumab + Gemcitabine + Cisplatin and 344 patients randomized to Placebo + Gemcitabine + Cisplatin (Full Analysis Set). Five of these patients did not receive treatment (resulting in 338 in Durvalumab arm and 342 in Placebo arm for Safety Analysis Set). Hence, the Total numbers at risk for all-cause mortality is 341 (Durvalumab) and 344 (Placebo), while the Total number at Risk by any Serious/Other Adverse Event is 338 (Durvalumab) and 342 (Placebo).
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Placebo + Gemcitabine + Cisplatin
All-Cause Mortality (participants affected / at risk) | 198/341 | 226/344
Serious Adverse Events (participants affected / at risk) | 160/338 | 149/342
Other Adverse Events (participants affected / at risk) | 326/338 | 330/342
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab + Gemcitabine + Cisplatin (N=338) | Placebo + Gemcitabine + Cisplatin (N=342)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Gastroenteritis escherichia coli (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella infection (Infections and infestations) | 0 (0) | 2 (2)
Liver abscess (Infections and infestations) | 1 (1) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 6 (7) | 7 (8)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 11 (11) | 9 (12)
Septic shock (Infections and infestations) | 1 (1) | 4 (6)
Urinary tract infection (Infections and infestations) | 6 (6) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chemical peritonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 4 (4)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (4) | 2 (2)
Platelet count decreased (Investigations) | 4 (4) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Immune-mediated arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 4 (4) | 1 (1)
Device malfunction (Product Issues) | 2 (2) | 2 (3)
Device occlusion (Product Issues) | 0 (0) | 4 (4)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Stent malfunction (Product Issues) | 0 (0) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 8 (11) | 4 (4)
Azotaemia (Renal and urinary disorders) | 1 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Angiopathy (Vascular disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 12 (16) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 8 (8)
Arterial thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 4 (5) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (6)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (3)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bicytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fistula of small intestine (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 3 (3) | 3 (3)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (3) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 5 (5)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Obstruction gastric (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (6) | 5 (5)
Asthenia (General disorders) | 1 (1) | 2 (2)
Death (General disorders) | 0 (0) | 2 (2)
Device related thrombosis (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 6 (6) | 4 (4)
Malaise (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 13 (16) | 8 (8)
Sudden death (General disorders) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 6 (8) | 7 (8)
Biloma rupture (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 25 (42) | 17 (20)
Cholangitis acute (Hepatobiliary disorders) | 4 (5) | 4 (7)
Cholecystitis (Hepatobiliary disorders) | 1 (3) | 4 (4)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder rupture (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cytolysis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 3 (3)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 1 (2) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 4 (4) | 5 (5)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess intestinal (Infections and infestations) | 1 (1) | 0 (0)
Acinetobacter sepsis (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 5 (5)
Biliary abscess (Infections and infestations) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 4 (4) | 2 (2)
Biliary tract infection (Infections and infestations) | 5 (7) | 7 (8)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Covid-19 (Infections and infestations) | 4 (4) | 2 (2)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Cholangitis infective (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 2 (3) | 3 (3)
Device related sepsis (Infections and infestations) | 1 (1) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 1 (1)
Gallbladder empyema (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab + Gemcitabine + Cisplatin (N=338) | Placebo + Gemcitabine + Cisplatin (N=342)
Urinary tract infection (Infections and infestations) | 18 (25) | 19 (20)
Alanine aminotransferase increased (Investigations) | 29 (37) | 34 (44)
Aspartate aminotransferase increased (Investigations) | 23 (30) | 31 (39)
Blood bilirubin increased (Investigations) | 9 (10) | 20 (22)
Blood creatinine increased (Investigations) | 10 (12) | 33 (43)
Gamma-glutamyltransferase increased (Investigations) | 12 (15) | 18 (27)
Neutrophil count decreased (Investigations) | 89 (225) | 105 (262)
Platelet count decreased (Investigations) | 68 (126) | 77 (175)
Weight decreased (Investigations) | 20 (20) | 20 (24)
White blood cell count decreased (Investigations) | 37 (78) | 46 (104)
Decreased appetite (Metabolism and nutrition disorders) | 85 (102) | 79 (91)
Hypokalaemia (Metabolism and nutrition disorders) | 28 (38) | 16 (24)
Hypomagnesaemia (Metabolism and nutrition disorders) | 32 (48) | 29 (34)
Hyponatraemia (Metabolism and nutrition disorders) | 22 (25) | 21 (23)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (22) | 14 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 28 (32) | 22 (24)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (20) | 19 (22)
Hypothyroidism (Endocrine disorders) | 22 (22) | 11 (11)
Dizziness (Nervous system disorders) | 21 (24) | 16 (20)
Dysgeusia (Nervous system disorders) | 20 (24) | 16 (22)
Headache (Nervous system disorders) | 23 (26) | 14 (18)
Insomnia (Psychiatric disorders) | 32 (34) | 36 (36)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (23) | 18 (18)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 (26) | 17 (20)
Alopecia (Skin and subcutaneous tissue disorders) | 28 (30) | 15 (15)
Pruritus (Skin and subcutaneous tissue disorders) | 38 (46) | 28 (30)
Rash (Skin and subcutaneous tissue disorders) | 38 (56) | 27 (34)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18 (21) | 8 (9)
Anaemia (Blood and lymphatic system disorders) | 159 (246) | 149 (246)
Abdominal pain (Gastrointestinal disorders) | 46 (59) | 54 (62)
Hypertension (Vascular disorders) | 19 (31) | 20 (23)
Abdominal pain upper (Gastrointestinal disorders) | 35 (41) | 30 (35)
Constipation (Gastrointestinal disorders) | 108 (133) | 99 (117)
Diarrhoea (Gastrointestinal disorders) | 54 (69) | 47 (74)
Dyspepsia (Gastrointestinal disorders) | 21 (24) | 25 (26)
Nausea (Gastrointestinal disorders) | 136 (211) | 117 (201)
Stomatitis (Gastrointestinal disorders) | 23 (29) | 22 (25)
Vomiting (Gastrointestinal disorders) | 59 (81) | 57 (84)
Leukopenia (Blood and lymphatic system disorders) | 20 (43) | 17 (34)
Asthenia (General disorders) | 47 (76) | 48 (70)
Fatigue (General disorders) | 87 (151) | 86 (123)
Oedema peripheral (General disorders) | 27 (31) | 17 (23)
Pyrexia (General disorders) | 60 (98) | 49 (84)
Neutropenia (Blood and lymphatic system disorders) | 106 (212) | 101 (204)
Thrombocytopenia (Blood and lymphatic system disorders) | 42 (67) | 42 (76)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT03875235/Prot_003.pdf
  • Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT03875235/SAP_004.pdf